CLINICAL TRIAL: NCT06986239
Title: Safety, Tolerability and Immunogenicity of One Single Administration of PCV-LITE, a Novel Adjuvanted Pneumococcal Conjugate Vaccine Supplemented With LiteVax Adjuvant, in Young Healthy Participants
Brief Title: Safety and Immunogenicity of PCV-LITE, a Low-dose of Pneumococcal Conjugate Vaccine With LiteVax Adjuvant
Acronym: PCV-LITE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: LiteVax BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-515972-11-00; 2024-515972-11-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-30; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Vaccine Reaction
Keywords: Vaccine adjuvant; LiteVax Adjuvant; Pneumococcal polysaccharide conjugate vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fractional dose of PCV20 (Experimental): A single intramuscular injection of 0.5 mL comprising 1/5th dose of Prevenar20 without LiteVax Adjuvant (LVA)
  Interventions: Biological: PCV-LITE
- Fractional dose of PCV20 plus LVA (Experimental): A single intramuscular injection of 0.5 mL comprising 1/5th dose of Prevenar20 with 1 mg of LiteVax Adjuvant (LVA)
  Interventions: Biological: PCV-LITE+LVA
- Standard dose of PCV20 without LVA (Active Comparator): A single intramuscular injection of 0.5 mL comprising a full dose of Prevenar20 without LiteVax Adjuvant
  Interventions: Biological: PCV20
- Standard dose of PCV20 plus 1 mg LiteVax Adjuvant (Experimental): A single intramuscular injection of 0.5 mL comprising a full dose of Prevenar20 with LiteVax Adjuvant
  Interventions: Biological: PCV20+LVA

INTERVENTIONS:
Biological: PCV-LITE — Fractional dose of pneumococcal polysaccharide conjugate vaccine without LiteVax Adjuvant (LVA)
  Arms: Fractional dose of PCV20
Biological: PCV-LITE+LVA — Fractional dose of pneumococcal polysaccharide conjugate vaccine with 1 mg of LiteVax Adjuvant (LVA)
  Arms: Fractional dose of PCV20 plus LVA
Biological: PCV20 — Standard (full) dose of pneumococcal polysaccharide conjugate vaccine without LiteVax Adjuvant (LVA)
  Arms: Standard dose of PCV20 without LVA
Biological: PCV20+LVA — Standard (full) dose of pneumococcal polysaccharide conjugate vaccine with LiteVax Adjuvant (LVA)
  Arms: Standard dose of PCV20 plus 1 mg LiteVax Adjuvant

SUMMARY:
Streptococcus pneumoniae is a common bacteria and major cause of serious infections like bloodstream infections, pneumonia, and meningitis. These infections are most common in children under 2 years old and adults over 65 years of age and dangerous for all age groups. Current vaccines, which contain parts of the bacteria, have significantly reduced the incidence of invasive pneumococcal disease (IPD). To broaden protection more serotypes are added to the vaccines over the years, which results in lower immune responses to the serotype-specific polysaccharides while a stronger vaccine is desired for older people and people with a weakened immune system. In addition, these complex vaccines are hardly affordable for the growing group of older adults in low- and middle-income countries (LMICs). To address these challenges, a new potent adjuvant called 'LiteVax Adjuvant' was developed. It has been shown to improve the efficacy of vaccines, even at low doses of antigen. A lower antigen dose reduces the costs of vaccines and promotes accessibility in LMICs. By testing a standard and a low dose of a commercial pneumococcal conjugate vaccine combined with LiteVax Adjuvant in healthy volunteers, we aim to determine whether the adjuvant enhances the immune response and if a lower vaccine dose is effective. At the same time, the safety of the vaccines is being investigated.

DETAILED DESCRIPTION:
The objectives are to evaluate the safety and the immunogenicity of a single intramuscular (IM) injection of a standard dose of PCV20 and a low dose of PCV20 (1/5th) with or without 1 mg of LVA immunoadjuvant.

This study is a randomized, Phase 1, single-center, observer-blind, active-controlled 4-arm study to evaluate the safety, tolerability, and immunogenicity of PCV-LITE, a novel adjuvanted pneumococcal conjugate vaccine. PCV-LITE consists of 1/5th-dose of PCV20 plus 1 mg of LVA (Cohort 2) and will be compared with 1/5th-dose of PCV20 without adjuvant (Cohort 1), a full dose of PCV20 plus 1 mg of LVA (Cohort 4) and a full dose of PCV20 without adjuvant (Cohort 3). The PCV20 will be the benchmark and the reference vaccine for the three study vaccines.

Cohort 1: 1/5th-dose of PCV20 (reference vaccine diluted in saline), Cohort 2: 1/5th-dose of PCV20 plus 1 mg LVA (study vaccine; PCV-LITE), Cohort 3: full dose of PCV20 (reference vaccine), and Cohort 4: full dose of PCV20 plus 1 mg LVA (study vaccine). A total of 80 participants are planned to be randomized, 20 per cohort. Dose increase of PCV20 (1/5th-dose to a full dose) occurs in two stages (N=40 in each stage). Two consecutive sentinel groups per dose level of PCV20 (first 4 participants on Day 1 followed by 6 participants on Day 4 after an uneventful 72-hours safety follow-up) are implemented to minimize risk to the participants. Participants will randomly be assigned in each stage. A screening visit, a baseline/vaccination visit and 3 follow-up visits at Day 8, Day 29 and Day 181 will be performed. Sentinels will have an additional follow-up telephone contact at Day 4. The study duration for each participant will be up to 21 days of screening, and 180 ± 15 days of follow-up after vaccination.

Participants will be healthy adults aged between 18 and 50 years (inclusive) who have had no laboratory confirmed S. pneumoniae infection in the 36 months prior to study vaccination and have not received an S. pneumoniae vaccination in the 36 months prior to study vaccination.

Interventions: All participants will receive one IM vaccination with the reference or study vaccine. The study vaccine will be prepared by an unblinded pharmacist and administered by an unblinded vaccinator while the participant and other site staff remain blinded (observer-blind). Solicited local and systemic AEs will be recorded in an electronic diary (eDiary) for 14 days after vaccination. The study team will closely monitor the eDiary during the 14-day follow-up period. At Day 15, the Investigator will review the data in the eDiary to determine whether an additional visit is required. If so, the participant should visit the site within 3 days. Unsolicited AEs will be monitored for 28 days after vaccination. SAEs, pIMDs and AESIs will be assessed for 180 days after vaccination. Blood samples (± 12 mL) will be collected from all participants at screening for eligibility evaluation and to examine haematology and biochemistry to check health status. Blood samples will be collected also at the other visits (maximal 20 mL/Visit, 4 visits). In order to evaluate whether the vaccines induce antibodies in the mucosa, mucosal nose swab samples of Mucosal Lining Fluid (MLF) will be collected from all participants at Visit 1/Day 1 and Visit 3/Day 29. The samples will be processed by a local lab (labelled, listed, and frozen) and analyzed by an external laboratory following qualified standard procedures.

ELIGIBILITY:
Inclusion Criteria:

* Written signed informed consent obtained before any study-related activities.
* Aged 18 to 50 years inclusive, at the time of signing the ICF.
* Participants who are considered to be in good general health as determined by medical evaluation including medical history, physical examination (PE) and laboratory tests within 21 days prior to enrolment.
* Participants with a BMI within the range 18.5 to 35 kg/m2 inclusive at screening.
* Women who are not pregnant or breastfeeding, and one of the following conditions applies:

  * Women of non-childbearing potential (WONCBP) OR
  * WOCBP and using a highly effective contraceptive method (with a failure rate of less than 1 % per year). Appendices from at least 1 month prior to study vaccination and for 3 months post-vaccination. The investigator should evaluate the potential for contraceptive method failure (e.g. noncompliance, recently initiated) in relationship to study vaccination. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the participant. The participant should commit to abstinence for at least 1 month prior to study vaccination and for 3 months post-vaccination. If the participant will not maintain abstinence and changes her status, the participant must first commit to another highly effective method of contraception, which should be discussed with the investigator prior to terminating sexual abstinence as contraceptive method.
* WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test before vaccination at Day 1. The investigator is responsible for review of medical history and menstrual history to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Participants who are willing and able to comply with the study procedures and are in the view of the investigator capable of completing the study.

Exclusion Criteria: Medical Conditions

* History of laboratory confirmed pneumococcal infection in the past 36 months prior to the day of study vaccination.
* Positive (in the past, suspected or ongoing) for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.
* Past or current history of immune-mediated and/or autoimmune diseases as indicated by the investigator, e.g. diabetes mellitus type I and thyroid disease.
* Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator.
* Clinical conditions representing a contraindication for IM administration, as judged by the investigator, e.g. history of bleeding disorder (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM administration or blood draws.
* History of confirmed hypersensitivity, allergy and/or anaphylaxis to diphtheria toxoid or to squalene-based adjuvants, or other components of the study vaccine (aluminum phosphate, succinic acid, Polysorbate 80).
* Current history of uncontrolled medical illness (unstable for the past 3 months) as judged by investigator, e.g. hypertension, diabetes mellitus type 2.
* Past or current history of any neurological disorder, e.g. Guillain-Barré syndrome and seizure disorder other than: 1) childhood febrile seizures, or 2) seizures that have not required treatment within the last 3 years.
* History of asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
* Active malignancy or malignancy within the past 5 years, except basocellular carcinoma (single lesion) that has been fully removed.
* Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past 2 years or that is expected to require the use of oral or intravenous corticosteroids.
* History of hereditary angioedema, acquired angioedema or idiopathic forms of angioedema.
* History of idiopathic urticaria within the past year.
* Current or recent (< 2 years ago) heavy smoking (> 20 cigarettes per day) or heavy vaping (> 2 mL e-liquid daily, which correspond with 20 cigarettes; reference ). If candidate stopped smoking or vaping > 2 years ago, the investigator would make an individual judgement based on the total packs or use per year and the candidate's overall health status. Drug - or alcohol abuse/addiction (including alcohol dependence), or psychiatric condition (e.g., past or present psychoses; disorder requiring lithium; or within 5 years prior to administration of study vaccine, a history of suicide plan or attempt), which in the investigator's opinion could compromise the participant's safety and/or compliance with the protocol.
* A rash, dermatological condition or tattoos that would, in the opinion of the investigator, interfere with injection local reaction rating.

Exclusion Criteria: Prior/Concomitant Therapy

* Prior receipt of an investigational or licensed pneumococcal vaccine in the 36 months before administration of study vaccine or planning to receive a pneumococcal vaccination during the study period.
* Prior receipt of a live attenuated vaccine in the 28 days prior to administration of study vaccine or within 14 days for subunit or inactivated vaccines other than pneumococcal vaccination.
* Planning to receive a vaccine during the first 28 days following the administration of study vaccine.
* Currently participating in another clinical study or planning to participate in another study during the study period, or administration of any investigational drug, vaccine or medical device in the 4 weeks prior to study vaccination.
* Prior receipt of blood, blood-derived products or immunoglobulins in the 6 months prior to administration of study vaccine or planning to receipt such product during the study period.
* Chronic administration (defined as 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to vaccination or planned administration during the study (excluding topical, inhaled and intranasal preparations and intra-articular injections). For corticosteroids, this is prednisone >= 20 mg/day, or equivalent.
* Current intake of more than 1 anticoagulant medication (coumarin derivatives, low molecular weight heparin, DOAC) or 1 anticoagulant medication in combination with anti-aggregation medication.
* Current anti-tuberculosis prophylaxis or therapy.
* Elective surgery planned in the first 14 days following study vaccination.

Exclusion Criteria:Others

* WOCBP who are pregnant, breast-feeding or planning to become pregnant during the study.
* Participants with history of any medical conditions that, in opinion of the investigator, might interfere with the results of the study or pose additional risk to the participants due to participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Solicited and non-solicited local and systemic adverse events after a single administration of Prevenar 20 with or without LiteVax adjuvant | Solicited AEs 14 days, non-solicited AEs 28 days and SAEs/pIMD/AESIs 180 days post-vaccination
  To evaluate the safety and tolerability of a single administration of 1/5th-dose of Prevenar 20 + 1 mg LVA (PCV-LITE), 1/5th-dose of Prevenar 20 without LVA, and a full-dose of Prevenar 20 + 1 mg LVA in comparison to a full-dose of Prevenar 20 without LVA, in healthy participants (18-50 years)
  * Occurrence of solicited local and systemic adverse events (AEs) for 14 days, unsolicited AEs for 28 days, and serious adverse events (SAEs), potential immune-mediated diseases (pIMDs), and adverse events of special interest (AESIs) for 180 days after vaccination.
  * Occurrence of clinically abnormal haematology and serum biochemistry laboratory values 1 day, 7 days, and 28 days, after vaccination versus baseline (Day 0, pre-vaccination).

SECONDARY OUTCOMES:
Humoral immune responses to a single administration of Prevenar 20 with or without LiteVax Adjuvant by multiplex immune assay (MIA) | Pre-vaccination (Day 0) and 28 and 180 days post-vaccination
  Humoral immune responses to low and full dose of Prevenar 20 with or without LiteVax Adjuvant (LVA) will be determined by a validated multiplex immune assay (MIA) in individual serum samples and expressed as arbitrary units. Geometric mean titers (GMTs), geometric mean concentrations (GMCs), standard deviation (SD), and 95% confidence intervals (95% CI) against the 20 vaccine serotypes will be calculated per cohort.
Humoral immune response to a single administration of Prevenar 20 with or without LiteVax Adjuvant measured by opsonophagocytic activity assay (OPA) | Pre-vaccination (Day 0), 28 days and optionally 180 days post-vaccination
  Humoral immune response to low and full dose of Prevenar 20 with or without LiteVax Adjuvant will be determined by a validated opsonophagocytic activity assay (OPA) in individual serum samples and expressed as arbitrary units. Geometric mean titers (GMTs), geometric mean concentrations (GMCs), standard deviations (SDs), and 95% confidence intervals (95% CIs) against the 20 vaccine serotypes or a selection thereof) will be calculated per cohort

OTHER OUTCOMES:
Functional serum antibody responses | Pre-vaccination (Day 0), and 28 and optionally 180 days post-vaccination and pre-vaccination
  Functional serum antibody responses to (a selection of) the 20 serotypes of PCV20 will be determined by validated .
Mucosal antibody response | Pre-vaccination (Day 0), and 28 days and optionally 180 days post-vaccination
  Mucosal (IgG and/or IgA) antibody titers in nasal swabs to (a selection of) the 20 serotypes of PCV20 will be determined by a validated multiplex immune assay (MIA) and expressed as arbitrary units.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Beek LF, van der Gaast-de Jongh C, Platenburg PP, Hilgers L, de Jonge MI. Improving the immunogenicity of the pneumococcal conjugate vaccine using a synthetic carbohydrate fatty acid monosulphate squalane-in-water adjuvant. Vaccine. 2025 Apr 2;51:126893. doi: 10.1016/j.vaccine.2025.126893. Epub 2025 Feb 20. PMID 39983540